CLINICAL TRIAL: NCT05640973
Title: Clinical Usability of a Novel Non-Adhesive Applicator for the Monitoring of tcPCO2 in Neonates
Brief Title: TCOM Ring Evaluation
Status: Withdrawn | Type: Observational
Why Stopped: Device was FDA approved before feasibility study could be performed
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Ann Donnelly, Principal Investigator, Milton S. Hershey Medical Center
Other Study IDs: 00020402
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Carbon Dioxide Partial Pressure Determination, Transcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation — Evaluation of ease of use

SUMMARY:
Subjects that are currently on a transcutaneous carbon dioxide monitor (TCOM) to monitor the carbon dioxide level in their blood will be placed on an additional TCOM using a non-adhesive sensor application ring instead of the usual adhesive ring to hold the TCOM sensor in place in order to evaluate usability of the non-adhesive applicator.

ELIGIBILITY:
Inclusion Criteria:

1. Premature or term birth newborn infants requiring transcutaneous monitoring
2. Thigh circumference of greater than 63mm
3. Weight greater than or equal to 600g
4. Ability of caretaker to understand verbal and written instructions and informed consent

Exclusion Criteria:

1. Absence of written informed consent.
2. Skin condition contraindicating transcutaneous measurements.
3. Thigh circumference less than or equal to 63 mm

Ages: 5 Minutes to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Usability of a Novel Non-Adhesive Applicator for the Monitoring of tcPCO2 in Neonates | 3 Months

IPD SHARING:
Plan to Share IPD: No